CLINICAL TRIAL: NCT06793215
Title: A Phase III, Randomized, Open-Label Study Evaluating the Efficacy and Safety of Divarasib and Pembrolizumab Versus Pembrolizumab and Pemetrexed and Carboplatin or Cisplatin in Patients With Previously Untreated, KRAS G12C-Mutated, Advanced or Metastatic Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study Evaluating the Efficacy and Safety of Divarasib and Pembrolizumab Versus Pembrolizumab and Pemetrexed and Carboplatin or Cisplatin in Participants With Previously Untreated, KRAS G12C-Mutated, Advanced or Metastatic Non-Squamous Non-Small Cell Lung Cancer
Acronym: Krascendo 2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO45042
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer; KRAS G12C Lung Cancer
Keywords: Advanced Non-Small Cell Lung Cancer; KRAS G12 Lung Cancer; Advanced Lung Cancer; Metastatic lung cancer; Divarasib; KRAS G12C Inhibitor; KRAS G12C Positive; KRAS Mutation; KRAS G12C Mutation; Lung Cancer Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pembrolizumab; Pemetrexed; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Divarasib + Pembrolizumab (Experimental): Participants will receive divarasib orally, once daily (QD) and pembrolizumab via intravenous (IV) infusion every 3 weeks (Q3W)
  Interventions: Drug: Divarasib; Drug: Pembrolizumab
- Pembrolizumab + Pemetrexed + Carboplatin or Cisplatin (Active Comparator): Participants will receive pembrolizumab, pemetrexed and carboplatin or cisplatin via IV infusion Q3W
  Interventions: Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin

INTERVENTIONS:
Drug: Divarasib — Divarasib will be administered orally QD
  Arms: Divarasib + Pembrolizumab
Drug: Pembrolizumab — Pembrolizumab will be administered via IV infusion Q3W
Drug: Pemetrexed — Pemetrexed will be administered via IV infusion Q3W
  Arms: Pembrolizumab + Pemetrexed + Carboplatin or Cisplatin
Drug: Carboplatin — Carboplatin will be administered via IV infusion Q3W
  Arms: Pembrolizumab + Pemetrexed + Carboplatin or Cisplatin
Drug: Cisplatin — Cisplatin will be administered via IV infusion Q3W
  Arms: Pembrolizumab + Pemetrexed + Carboplatin or Cisplatin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of divarasib and pembrolizumab compared with pembrolizumab and pemetrexed and carboplatin or cisplatin, for the first-line treatment of adult participants with KRAS G12C-mutated, advanced or metastatic non squamous non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically or cytologically confirmed diagnosis of advanced or metastatic non squamous NSCLC that is not eligible for curative surgery and/or definitive chemoradiotherapy
* Measurable disease, as defined by RECIST v1.1
* No prior systemic treatment for advanced or metastatic NSCLC
* Documentation of the presence of a KRAS G12C mutation
* Documentation of known PD-L1 expression status in tumor tissue
* Availability of a representative tumor specimen
* Adequate end-organ function
* Eligible to receive a platinum-based chemotherapy regimen

Exclusion Criteria Related to NSCLC:

* Known concomitant second oncogenic driver with available targeted treatment
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for >=2 weeks prior to randomization
* History of leptomeningeal disease
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once a month or more frequently)

Exclusion Criteria Related to Current or Prior Treatments:

* Any anti-cancer systemic therapy, including hormonal therapy, within 21 days prior to randomization, or is expected to require any other form of antineoplastic therapy while in the study
* Radiation therapy including palliative RT to bone metastases within 2 weeks prior to randomization and RT to the lung >30Gy within 6 months prior to randomization
* Prior treatment with KRAS G12C inhibitors or pan-KRAS/RAS inhibitors
* Treatment with systemic immunosuppressive or immunostimulatory medications, including CD137 agonists and immune checkpoint inhibitors
* Current treatment with medications that are well known to prolong the QT interval
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to randomization
* Prior allogeneic stem cell or solid organ transplantation

Exclusion Criteria Related to General Health:

* History of malignancy other than NSCLC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year overall survival [OS] rate >90%), such as adequately treated carcinoma in situ of the cervix, non melanoma skin carcinoma, localized prostate cancer, ductal breast carcinoma in situ, or Stage I uterine cancer
* Individuals with chronic diarrhea, short bowel syndrome or significant upper gastrointestinal surgery including gastric resection, a history of inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis) or any active bowel inflammation (including diverticulitis), malabsorption syndrome, conditions that would interfere with enteral absorption
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on the screening chest computed tomography scan
* Significant cardiovascular disease within 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 5 years
  PFS is defined as the time from randomization to the first occurrence of disease progression, as determined by blinded independent central review (BICR) according to RECIST v1.1, or death from any cause (whichever occurs first)
Overall Survival (OS) | Up to approximately 5 years
  OS is defined as the time from randomization to death from any cause

SECONDARY OUTCOMES:
Objective Response | Up to approximately 5 years
  Objective response is defined as complete response (CR) or partial response (PR) on two consecutive occasions >=4 weeks apart, as determined by BICR according to RECIST v1.1
Change from Baseline on the European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire-Supplemental Lung Cancer Module (EORTC QLQ-LC13) Cough Scale | Baseline up to Cycle 5 Day 1 (each cycle is 21 days)
Change from Baseline on the EORTC Quality of Life Questionnaire (QLQ-C30) Dyspnea Item and Physical Functioning Scale | Baseline up to Cycle 5 Day 1 (each cycle is 21 days)
Duration of Response (DOR) | Up to approximately 5 years
  DOR is defined as the time from the first occurrence of a documented objective response to disease progression, as determined by BICR according to RECIST v1.1, or death from any cause (whichever occurs first)
Percentage of Participants with Adverse Events (AEs) | Up to approximately 5 years
Number of Participants Reporting Presence, Frequency, Severity, and/or Degree of Interference with Daily Function of Symptomatic Treatment Toxicities Assessed by NCI Patient-Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to approximately 5 years
Change from Baseline in the Severity of Selected Symptomatic Treatment Toxicities as Assessed Through use of the NCI PRO-CTCAE | Up to approximately 5 years
Frequency of Participants' Response of the Degree they are Troubled with Treatment Symptoms, as Assessed Through use of the single-item EORTC Item List (IL46) | Up to approximately 5 years
Change from Baseline on the EORTC QLQ-C30 and QLQ-LC13 Functional and Global Health Status Score/Quality of Life Score (GHS/QoL) | Up to approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (151):
- United States (21):
  - Alaska Oncology and Hematology, Anchorage, Alaska
  - Marin Cancer Care Inc, Greenbrae, California
  - BioResearch Partner, Hialeah, Florida
  - Piedmont Cancer Institute, PC, Atlanta, Georgia
  - Summit Cancer Care PC, Savannah, Georgia
  - St. Luke's Cancer Institute, Boise, Idaho
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - Profound Research, LLC, Farmington Hills, Michigan
  - Missouri Baptist Medical Center, St Louis, Missouri
  - San Juan Oncology Associates, Farmington, New Mexico
  - Montefiore Einstein Cancer Center, The Bronx, New York
  - Clinical Research Alliance, Westbury, New York
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Baptist Cancer Center, Memphis, Tennessee
  - Renovatio Clinical - El Paso, El Paso, Texas
  - JPS Health Network, Fort Worth, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Community Clinical Trials, Kingwood, Texas
  - Texas Tech Health Science Center, Lubbock, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - University of Texas Health Center at Tyler, Tyler, Texas
- Argentina (2):
  - Hospital Britanico, Ciudad Autonoma Buenos Aires
  - Centro Oncologico Korben, Ciudad Autonoma Buenos Aires
- Australia (6):
  - Kinghorn Cancer Centre, Darlinghurst, New South Wales
  - Calvary Mater Newcastle, Warath, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
- Belgium (4):
  - AZORG Campus Aalst-Moorselbaan, Aalst
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - CHU HELORA - Hôpital de Mons - Site Kennedy, Mons
  - AZ Delta (Campus Rumbeke), Roeselare
- Brazil (7):
  - Crio - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Centro Integrado de Oncologia de Curitiba, Curitiba, Paraná
  - Liga Norte Riograndense Contra O Câncer, Natal, Rio Grande do Norte
  - Irmandade Da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII Hospital de Câncer de Barretos, Barretos, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
- Canada (4):
  - BC Cancer ? Kelowna (Sindi Ahluwalia Hawkins Centre), Kelowna, British Columbia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Centre Hospitalier Regional De Rimouski, Rimouski, Quebec
- China (4):
  - West China Hospital - Sichuan University, Chengdu
  - Sir Run Run Shaw Hospital Zhejiang University, Hangzhou
  - Shanghai Pulmonary Hospital, Shanghai
  - Shanghai East Hospital, Shanghai
- Denmark (4):
  - Aarhus Universitetshospital, Aarhus N
  - Herlev Hospital, Afdeling for Kræftbehandling, Center for Kræftforskning, Klinisk Forskningsenhed, Herlev
  - Rigshospitalet, København Ø
  - Sjællands Universitetshospital, Roskilde, Roskilde
- France (12):
  - CHU Angers, Angers
  - Hopital Avicenne, Bobigny
  - Hôpital Louis Pradel, Hospices Civils de Lyon, Bron
  - Centre Francois Baclesse, Caen
  - Centre Leon Berard, Lyon
  - CHU Montpellier, Montpellier
  - Groupe Hospitalier Paris Saint Joseph, Paris
  - Hopital Tenon, Paris
  - CHU Bordeaux, Pessac
  - Centre Hospitalier Universitaire de Reims, Reims
  - CH de Saint Quentin, Saint-Quentin
  - Centre Hospitalier Bretagne Atlantique Vannes, Vannes
- Germany (17):
  - Vivantes - Klinikum Im Friedrichshain;Innere Medizin ? Hämatologie, Onkologie und Palliativmedizin, Berlin
  - Charite - Universitätsmedizin Berlin, Berlin
  - Technische Universität Dresden - Medizinische Fakultät Carl Gustav Carus;Medizinische Klinik und Poliklinik I, Dresden
  - KEM/Evang. Kliniken Essen Mitte gGmbH, Essen
  - Universitätsklinikum Essen, Essen
  - Klinikum Esslingen, Esslingen am Neckar
  - Asklepios Fachkliniken GmbH, Gauting
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - KRH Klinikum Siloah-Oststadt-Heidehaus, Hanover
  - Universität Des Saarlandes, Homburg
  - Lungenfachklinik Immenhausen, Immenhausen
  - Vincentius-Diakonissen-Kliniken gAG, Karlsruhe
  - SLK Kliniken Heilbronn GmbH, Standort Fachklinik Löwenstein, Löwenstein
  - Universität Mannheim, Mannheim
  - Pius Hospital Oldenburg, Oldenburg
  - Universitätsklinikum Regensburg, Regensburg
- Greece (4):
  - Alexandras Hospital, Athens
  - Errikos Dynan Hospital, Athens
  - Interbalkan Medical Center of Thessaloniki, Thessaloniki
  - Ag. Loukas Hospital, Thessaloniki
- Hong Kong (4):
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
  - Queen Elizabeth Hospital Department of Clinical Oncology, Kowloon
  - Prince of Wales Hosp, Shatin
- Hungary (2):
  - Matrai Gyogyintezet, Mátraháza
  - Reformatus Pulmonologiai Centrum, Törökbálint
- Italy (6):
  - Ospedale Giuseppe Moscati, Statte, Apulia
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Campania
  - Presidio san salvatore muraglia, Pesaro, Emilia-Romagna
  - IEO Istituto Europeo di Oncologia, Milan, Lombardy
  - USL 6 Toscana Nord Ovest ? P.O. Livorno, Livorno, Tuscany
  - Ospedale P. Pederzoli Casa di cura Privata, Peschiera Del Garda (VR), Veneto
- The Cancer Institute Hospital of JFCR, Tokyo, Japan
- Netherlands (3):
  - Amphia Ziekenhuis, Breda
  - Ziekenhuis St. Jansdal, Harderwijk
  - Isala, Zwolle
- Harbour Cancer and Wellness, Auckland, New Zealand
- Poland (10):
  - Centrum Pulmonologii i Torakochirurgii, Bystra
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Krakowski Szpital Specjalistyczny im sw.Jana Pawla II, Krakow
  - Uniwersytecki Szpital Kliniczny nr 4 w Lublinie, Lublin
  - Warminsko-Mazurskie Centrum Chorób P?uc w Olsztynie, Olsztyn
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii w Poznaniu, Poznan
  - Radomskie Centrum Onkologii, Radom
  - Instytut Gruzlicy I Chorob Pluc, Warsaw
  - Mazowiecki Szpital Onkologiczny, Wieliszew
  - Dolnoslaskie Centrum Chorob Pluc, Wroclaw
- Portugal (4):
  - Hospital de Braga, Braga
  - Hospital Beatriz Angelo, Loures
  - IPO do Porto, Porto
  - CHVNG/E_Unidade 1, Vila Nova de Gaia
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
- South Korea (6):
  - Pusan National University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Chilgok Hospital, Daegu
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (10):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Clinica Universidad de Navarra Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
- Switzerland (3):
  - Universitaetsspital Basel, Basel
  - Kantonsspital Graubünden Medizin Onkologie, Chur
  - Hôpital Universitaire de Genève (HUG), Geneva
- Taiwan (7):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-DA Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Cancer Center, Zhongzheng Dist.
- United Kingdom (7):
  - Blackpool Teaching Hospitals NHS Foundation Trust , Victoria Hospital, Blackpool
  - Bristol Haematology & Oncology Centre, Bristol
  - East Kent Hospitals University NHS Foundation Trust, Canterbury
  - Velindre NHS Trust - Velindre Cancer Centre, Cardiff
  - Barts and the London NHS Trust, London
  - Royal Marsden Hospital - Fulham, London
  - Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing